CLINICAL TRIAL: NCT03916159
Title: Extrauterine Placental Transfusion In Neonatal Resuscitation (EXPLAIN) of Very Low Birth Weight Infants (VLBW): A Randomized Clinical Trial
Brief Title: Extrauterine Placental Transfusion In Neonatal Resuscitation Of Very Low Birth Weight Infants
Acronym: EXPLAIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Köln (Other)
Responsible Party: Principal Investigator, Andre Oberthür, Principal Investigator, Universitätsklinikum Köln
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 18-232; DRKS00017041 (Registry Identifier: German Clinical Trials Register)
Record Dates: First submitted 2019-04-05; First posted 2019-04-16 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Very Low Birth Weight Infant; Placental Transfusion; Anemia
Keywords: extrauterine placental transfusion; delayed cord clamping; neonatal resuscitation
MeSH Terms: conditions — Fetofetal Transfusion; Anemia | interventions — Umbilical Cord Clamping; Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Extrauterine Placental Transfusion EPT (Experimental): Intervention group
  Interventions: Procedure: Extrauterine placental transfusion (Intervention group)
- Delayed cord clamping DCC (Active Comparator): Control group
  Interventions: Procedure: Delayed cord clamping (Control group)

INTERVENTIONS:
Procedure: Extrauterine placental transfusion (Intervention group) — At delivery by caesarean section, the infant is born with the placenta still attached via the umbilical cord and placental transfusion is performed at least 1 minute but not more than 10 minutes by holding the placenta ~40-50cm above the babies' heart level while respiratory support by mask continuous-positive-airway-pressure (CPAP) is initiated simultaneously.
  Arms: Extrauterine Placental Transfusion EPT
Procedure: Delayed cord clamping (Control group) — At delivery by caesarean section, delayed cord clamping will be performed by having the delivering obstetrician delay clamping of the umbilical cord for at least 30 seconds with initiation of respiratory support by mask CPAP after cord clamping.
  Arms: Delayed cord clamping DCC

SUMMARY:
To investigate the effect of extrauterine placental transfusion (EPT) compared to delayed cord clamping (DCC) on the mean hematokrit on the first day of life in very low birth weight infants (VLBW) born by caesarian section. The investigators hypothesize that EPT provides higher blood volume during neonatal transition and improves neonatal outcome of VLBW infants.

DETAILED DESCRIPTION:
This prospective randomized controlled study will be conducted among 2 groups, all of them are preterm infants with birth weight less than 1500 g ("very low birth weight" (VLBW)) who are delivered by caesarean section, in the first interventional group an extrauterine placental transfusion (EPT) will be done during neonatal resuscitation with respiratory pressure support. There will be a delayed cord clamping (DCC) of at least 30 - 60 seconds in the control group, before starting neonatal resuscitation with respiratory support.

In EPT approach preterm born infants are delivered by caesarean section with the placenta still attached to the infant via the umbilical cord. Then, placental transfusion is performed up to several minutes by holding the placenta ~40-50cm above the babies' heart level while respiratory support by mask continuous-positive-airway-pressure (CPAP) is initiated simultaneously.

Extrauterine placental transfusion may give more blood in babies delivered by cesarean section and may improve perfusion during the fetal-to-neonatal transition with impact on neonatal outcome.

ELIGIBILITY:
Inclusion Criteria:

* Birth weight < 1500 gram ("very low birth weight infant")
* Delivery by caesarean section
* Gestational age > 23+6 weeks

Exclusion Criteria:

* Vaginal delivery
* Fetal or maternal risk (i.e. compromise, emergency c-section)
* Congenital anomalies and/or major cardiac defects
* Placental abruption or previa with hemorrhage
* Placenta accreta or increta
* Monochorionic multiples (i.e. Di/Mo or Mo/Mo twins)
* Parents declined study

Min Age: 24 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2021-12-05 (Actual); Study Completion 2023-10-24 (Actual)

PRIMARY OUTCOMES:
Hematocrit | 0 - 24 hours of life
  Mean Hematocrit in the first 24 hours of life

SECONDARY OUTCOMES:
Cerebral tissue oxygen saturation | During first hour of life
  Transcutaneous measured cerebral tissue oxygen saturation given in percent (%) during neonatal resuscitation
Mean airway pressure | During first hour of life
  Mean airway pressure given in cmH2O during neonatal resuscitation
Mean tidal volume | During first hour of life
  Mean tidal volume given in milliliter (ml) during neonatal resuscitation
Heart rate | During first hour of life
  Heart rate given in beats-per-minute (bpm) during neonatal resuscitation
Blood oxygen saturation | During first hour of life
  Transcutaneous measured blood oxygen saturation given in percent (%) during neonatal resuscitation
Admission temperature | Admission to ward is up to 120 minutes of age
  Mean temperature at admission
All Grade Intraventricular Hemorrhage (IVH) | Up to 28 days of life
  Incidence of any intraventricular hemorrhage (grades 1-4)
All Grade BPD | At the corrected age of 36 weeks
  Incidence of Bronchopulmonary Disease (BPD) (all grades)
Spontaneous Pneumothorax/Pneumoperitoneum | During the first 7 days of life
  Early incidence of spontaneous pneumothorax and/or pneumoperitoneum
Spontaneous Pneumothorax/Pneumoperitoneum | Between day 7 and day 28 of life
  Late incidence of spontaneous pneumothorax and/or pneumoperitoneum
NEC/SIP with surgery | During the first 28 days of life
  Incidence of necrotizing enterocolitis (NEC) and/or spontaneous intestinal perforation (SIP) with need for surgery
Retinopathy of Prematurity (ROP), higher grades | At the corrected age of 40 weeks
  Incidence of retinopathy of prematurity with treatment (drugs and/or surgery)
Death | Until corrected age of 40 weeks
  Incidence of death in studied infants
Number of participants who received red blood cell (RBC) transfusion | During the first 7 days of life
  Amount of RBC Transfusion [cumulative ml/kg over the first 7 days] in those participants who received RBC transfusion
Hyperbilirubinemia | During the first 14 days of life
  Peak bilirubin concentration
Blood Exchange Transfusion | During the first 14 days of life
  Incidence of blood exchange transfusion due to critical hyperbilirubinemia of the neonate.
Intubation and Mechanical Ventilation | During the first 72 hours of life
  Incidence of intubation and time duration of mechanical ventilation
Intubation and Mechanical Ventilation | During hospitalization
  Incidence of intubation and time duration of mechanical ventilation
Neurodevelopmental Outcome | 22-26 month corrected gestational age
  Bayley Scales of Infant and Toddler Development - Third Edition (Bayley-III) composite score (motor, cognitive, language)

CONTACTS AND LOCATIONS:
Overall Officials: André Oberthuer, MD, Principal Investigator — University hospital of Cologne, Department of Pediatrics
Locations (1):
- University Hospital of Cologne, Department of pediatrics, Cologne, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kuehne B, Kirchgaessner C, Becker I, Kuckelkorn M, Valter M, Kribs A, Oberthuer A. Mask Continuous Positive Airway Pressure Therapy with Simultaneous Extrauterine Placental Transfusion for Resuscitation of Preterm Infants - A Preliminary Study. Biomed Hub. 2018 Jun 26;3(2):1-10. doi: 10.1159/000488926. eCollection 2018 May-Aug. PMID 31988958
- [Result] Kuehne B, Gruttner B, Hellmich M, Hero B, Kribs A, Oberthuer A. Extrauterine Placental Perfusion and Oxygenation in Infants With Very Low Birth Weight: A Randomized Clinical Trial. JAMA Netw Open. 2023 Nov 1;6(11):e2340597. doi: 10.1001/jamanetworkopen.2023.40597. PMID 37921769
- [Derived] Kuehne B, Hellmich M, Heine E, Kribs A, Mehler K, Oberthuer A. Neurodevelopmental Outcomes of Very Low Birth Weight Infants Following Extrauterine Placental Perfusion: A Follow-Up Study. Acta Paediatr. 2025 Sep;114(9):2246-2252. doi: 10.1111/apa.70101. Epub 2025 Apr 18. PMID 40251781